CLINICAL TRIAL: NCT05961514
Title: The Randomized Controlled Trial of Prostate Cancer Screening in Beijing, China
Brief Title: the Beijing Randomized Study Of Prostate Cancer Screening
Acronym: BROPCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022-1G-1021
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; MRI; Biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional (Other): The traditional/control arm consists of systematic biopsies of the prostate if PSA>4ng/ml.
  Interventions: Diagnostic Test: systemic biopsies
- Experimental (Experimental): The experimental arm consists of MRI tests and targeted biopsies if PI-RADS scores ≥3 or systematic biopsies if PSA>10ng/ml.
  Interventions: Diagnostic Test: Target biopsies

INTERVENTIONS:
Diagnostic Test: Target biopsies — MRI/Fusion target biopsies combine magnetic resonance imaging (MRI) with ultrasound-guided biopsy techniques to obtain tissue samples from areas of the prostate gland that appear abnormal on MRI.
  Arms: Experimental
Diagnostic Test: systemic biopsies — transrectal ultrasound (TRUS) guided prostate systemic biopsies
  Arms: Traditional

SUMMARY:
BROPCS is a randomized trial study comparing the effectiveness of traditional systematic biopsies and bpMRI followed targeted biopsies with PSA > 4ng/ml in initial screening.

DETAILED DESCRIPTION:
The aim of BROPCS study is to explore a suitable prostate cancer screening model for Chinese population, which can increase the specificity in early detection of prostate cancer without decreasing the sensitivity of clinically significant prostate cancers, and can reduce prostate cancer-specific mortality.This study will use a cluster randomized controlled trial method with a total of approximately 30,000 participants. The subjects will be randomly assigned to a control group (about 20,000 people) and a screening group (about 10,000 people), and some basic information will be obtained through a questionnaire survey. The screening group will undergo initial prostate-specific antigen (PSA) screening, and high-risk subjects (PSA > 4ng/ml) will be randomly assigned to two groups. The standard biopsy group will undergo traditional systematic biopsy, while the precision screening group will undergo further MRI examination and targeted fusion biopsy for those with positive MRI results.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men aged 60-75 with a life expectancy of more than 10 years;
2. Residing continuously in the community for more than 3 years and not previously diagnosed with prostate cancer;
3. Willing to participate in this project.

Exclusion Criteria:

1. Previously diagnosed with prostate cancer;
2. Previously diagnosed with any malignant tumor within the past 5 years;
3. Used medication within the past 3 months that can affect PSA values, mainly finasteride, dutasteride, and ketoconazole;
4. Recently had acute prostatitis, acute urinary retention, or underwent transurethral procedures (such as urethral dilation, urinary catheterization, cystoscopy, etc.) within the past week;
5. Have other serious illnesses or cannot perform activities of daily living independently.

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30000 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
detection of clinically significant prostate cancer （Gleason Score ≥7） | At 2 months after the last included biopsy procedure
  Cancers detected by pathological evaluation of biopsy specimen collected from the respective study arm

SECONDARY OUTCOMES:
detection of clinically insignificant prostate cancer （Gleason Score 3+3） | At 2 months after the last included biopsy procedure
  Cancers detected by pathological evaluation of biopsy specimen collected from the respective study arm

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital &institute, Beijing, Beijing Municipality, China